CLINICAL TRIAL: NCT01185353
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Parallel-Group, Phase 2b Study of LY3009104 in Patients With Active Rheumatoid Arthritis on Background Methotrexate Therapy
Brief Title: A Study in Participants With Rheumatoid Arthritis on Background Methotrexate Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13854; I4V-MC-JADA (Other: Eli Lilly and Company); CTRI/2011/06/001834 (Registry Identifier: Clinical Trials Registry India)
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-05

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib; Janus Kinases; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 mg LY3009104 once daily (Experimental): Administered orally once daily for initial 12 weeks followed by randomization to either 4 mg LY3009104 once daily or 2 mg LY3009104 twice daily for an additional 12 weeks. After 24 weeks of treatment participants will be eligible to participate in an open-label extension period (Part C). Part C: 4 mg or 8 mg administered orally once daily for 52 additional weeks. After 76 weeks of treatment participants will be eligible to participate in an additional open-label extension period (Part D). Part D: 4 mg administered orally once daily for 52 additional weeks.
  Interventions: Drug: LY3009104; Drug: Methotrexate
- 2 mg LY3009104 once daily (Experimental): Administered orally once daily for 24 weeks. After 24 weeks of treatment participants will be eligible to participate in an open-label extension period (Part C). Part C: 4 mg or 8 mg administered orally once daily for 52 additional weeks. After 76 weeks of treatment participants will be eligible to participate in an additional open-label extension period (Part D). Part D: 4 mg administered orally once daily for 52 additional weeks.
  Interventions: Drug: LY3009104; Drug: Methotrexate
- 4 mg LY3009104 once daily (Experimental): Administered orally once daily for 24 weeks. After 24 weeks of treatment participants will be eligible to participate in an open-label extension period (Part C). Part C: 4 mg or 8 mg administered orally once daily for 52 additional weeks. After 76 weeks of treatment participants will be eligible to participate in an additional open-label extension period (Part D). Part D: 4 mg administered orally once daily for 52 additional weeks.
  Interventions: Drug: LY3009104; Drug: Methotrexate
- 8 mg LY3009104 once daily (Experimental): Administered orally once daily for 24 weeks. After 24 weeks of treatment participants will be eligible to participate in an open-label extension period (Part C). Part C: 8 mg administered orally once daily for 52 additional weeks. After 76 weeks of treatment participants will be eligible to participate in an additional open-label extension period (Part D). Part D: 4 mg administered orally once daily for 52 additional weeks.
  Interventions: Drug: LY3009104; Drug: Methotrexate
- Placebo once daily (Placebo Comparator): Placebo administered orally once daily for initial 12 weeks followed by randomization to either 4 mg LY3009104 once daily or 2 mg LY3009104 twice daily for an additional 12 weeks. After 24 weeks of treatment participants will be eligible to participate in an open-label extension period (Part C). Part C: 4 mg or 8 mg administered orally once daily for 52 additional weeks. After 76 weeks of treatment participants will be eligible to participate in an additional open-label extension period (Part D). Part D: 4 mg administered orally once daily for 52 additional weeks.
  Interventions: Drug: Placebo; Drug: Methotrexate
- 2 mg LY3009104 twice daily (Experimental): (Not utilized in Part A) After 12 weeks treatment with 1 mg LY3009104 once daily or Placebo once daily in Part A, administered orally twice daily for 12 weeks. After 24 weeks of treatment participants will be eligible to participate in an open-label extension period (Part C). Part C: 4 mg or 8 mg administered orally once daily for 52 additional weeks. After 76 weeks of treatment participants will be eligible to participate in an additional open-label extension period (Part D). Part D: 4 mg administered orally once daily for 52 additional weeks.
  Interventions: Drug: LY3009104; Drug: Methotrexate

INTERVENTIONS:
Drug: LY3009104 — Administered orally
  Other Names: Janus Kinase (JAK)1/JAK2 Inhibitor; JAK1/2 Inhibitor; INCB028050; baricitinib
  Arms: 1 mg LY3009104 once daily; 2 mg LY3009104 once daily; 2 mg LY3009104 twice daily; 4 mg LY3009104 once daily; 8 mg LY3009104 once daily
Drug: Placebo — Administered orally
  Arms: Placebo once daily
Drug: Methotrexate — Administered orally as background therapy

SUMMARY:
The purpose of this trial is to evaluate the safety and efficacy of LY3009104 in participants with Rheumatoid Arthritis (RA).

DETAILED DESCRIPTION:
This study consists of the following:

* Screening period: 4 to 28-days
* Part A: a 12-week blinded, placebo controlled treatment period
* Part B: a 12-week blinded extension period
* Part C: an optional 52-week open-label extension period
* Part D: an additional optional 52-week open-label extension period
* Follow up period: 28 days

ELIGIBILITY:
Inclusion Criteria:

* Must have active RA
* Must regularly use methotrexate (MTX) for at least 12 weeks before your participation in this study
* Must have American College of Rheumatology (ACR) functional class I, II, or III
* Must have C-reactive protein (CRP) measurement > 1.2 times upper limit of normal (ULN) or Erythrocyte Sedimentation Rate (ESR) > ULN [28 millimeters/hour (mm/hr)]
* Have laboratory values that in the opinion of the investigator do not pose an unacceptable risk to the participants if study drug would be administered
* Must have venous access sufficient to allow blood sampling as per the protocol
* Must be reliable and willing to be available for the duration of the study and are willing to follow study procedures
* Must be able to read, understand, and give written informed consent approved by Lilly or its designee and the ethical review board (ERB) governing the site
* Male participants: agree to use 2 forms of highly effective methods of birth control with female partners of childbearing potential during the study
* If you are a woman and you could become pregnant during this study, you must talk to the study doctor about birth control. You are required to use 2 forms of highly effective methods of birth control to avoid getting pregnant during the study
* If you are a post-menopausal woman, you must be at least 45 years of age and have not menstruated for the last 12 months
* If you are a woman between 40 and 45 years of age, test negative for pregnancy, and have not menstruated during the last 12 months only, you must have an additional blood test
* For participants receiving corticosteroids, you must be on a dose not to exceed 10 mg of prednisone daily (or equivalent) and have been on the same dosing regimen for at least 6 weeks prior to randomization
* Continue to meet inclusion criteria for Parts A and B as applicable
* Part D only: have completed the 52 weeks (Week 24 to Week 76) of participation in Part C of the study without permanent study drug discontinuation and have not completed the Follow-Up Visit (approximately 28 days after the last dose of study drug)

Exclusion Criteria:

* Must not have received any parenteral corticosteroid administered by intra-articular, intramuscular (IM), or intravenous (IV) injection within 6 weeks prior to baseline
* Must not be concomitantly using non-steroidal anti-inflammatory drugs (NSAIDS), unless you are on a stable dose within the last 4 weeks
* Must not have received any prior biologic disease modifying anti-rheumatic drug (DMARD) therapy [such as Tumor necrosis factor-alpha (TNFα), interleukin (IL)-1, IL-6, T-cell or B-cell target therapies)
* Must not have used DMARDs other than methotrexate (MTX), hydroxychloroquine, or sulfasalazine within the last 8 weeks
* Must not have used leflunomide within the last 12 weeks and have not received cholestyramine to speed up the elimination of leflunomide from your body
* Must not have previously been randomized, completed or withdrawn from this study or any other study investigating LY3009104
* Must not have received prior treatment with an oral JAK inhibitor
* Must not have a current or recent (within the last 30 days) viral, bacterial, fungal, or parasitic infection
* Must not have had a serious infection (for example, pneumonia, cellulitis, or bone or joint infections) or atypical mycobacterial infection within the last 6 months
* Must not have had symptomatic herpes zoster or herpes simplex infection within the last 90 days or have a history of disseminated/complicated herpes zoster
* Must not have evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies
* Must not have evidence of hepatitis C virus (HCV) or active hepatitis B
* Must not have evidence or suspicion of active or latent tuberculosis (TB)
* Must not have another serious disorder or illness
* Must not be exposed to a live vaccine within the last 12 weeks
* Must not have donated more than 500 milliliters (mL) of blood within the last month
* Must not have had surgery on a joint that is to be assessed in the study within the last 2 months, or will require such during the study
* Must not be currently enrolled in, or discontinued within the last 30 days from a clinical trial involving an investigational drug or device or off-label use of a drug, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Presence of significant uncontrolled cerebro-cardiovascular [for example (eg), myocardial infarction (MI), unstable angina (UA), unstable arterial hypertension, severe heart failure or cerebrovascular accident], respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematologic or neuropsychiatric disorders, or abnormal laboratory values that in the opinion of the investigator pose an unacceptable risk to the participant if study drug would be administered

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (68):
- United States (31):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paradise Valley, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Covina, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Maria, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westlake Village, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aventura, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boca Raton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jupiter, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Mary, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Naples, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Harbor, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vero Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Bend, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flowood, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lincoln, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freehold, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Success, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middleburg Heights, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duncansville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
- Croatia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osijek
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb
- Czechia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Česká Lípa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hlučín
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hostivice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hustopeče
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zlín
- Hungary (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kistarcsa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Veszprém
- India (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahmedabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trivandrum
- Mexico (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cuauhtémoc
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., León
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Częstochowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Romania (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bacau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Galati
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
- Ukraine (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiev
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Simferopol
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ternopil
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vinnytsia

REFERENCES:
- [Derived] Taylor PC, Takeuchi T, Burmester GR, Durez P, Smolen JS, Deberdt W, Issa M, Terres JR, Bello N, Winthrop KL. Safety of baricitinib for the treatment of rheumatoid arthritis over a median of 4.6 and up to 9.3 years of treatment: final results from long-term extension study and integrated database. Ann Rheum Dis. 2022 Mar;81(3):335-343. doi: 10.1136/annrheumdis-2021-221276. Epub 2021 Oct 27. PMID 34706874
- [Derived] Combe B, Balsa A, Sarzi-Puttini P, Tony HP, de la Torre I, Rogai V, Durand F, Witt S, Zhong J, Dougados M. Efficacy and safety data based on historical or pre-existing conditions at baseline for patients with active rheumatoid arthritis who were treated with baricitinib. Ann Rheum Dis. 2019 Aug;78(8):1135-1138. doi: 10.1136/annrheumdis-2018-214261. Epub 2019 Mar 6. No abstract available. PMID 30842122
- [Derived] Peterfy C, DiCarlo J, Emery P, Genovese MC, Keystone EC, Taylor PC, Schlichting DE, Beattie SD, Luchi M, Macias W. MRI and Dose Selection in a Phase II Trial of Baricitinib with Conventional Synthetic Disease-modifying Antirheumatic Drugs in Rheumatoid Arthritis. J Rheumatol. 2019 Aug;46(8):887-895. doi: 10.3899/jrheum.171469. Epub 2019 Jan 15. PMID 30647190
- [Derived] Taylor PC, Kremer JM, Emery P, Zuckerman SH, Ruotolo G, Zhong J, Chen L, Witt S, Saifan C, Kurzawa M, Otvos JD, Connelly MA, Macias WL, Schlichting DE, Rooney TP, de Bono S, McInnes IB. Lipid profile and effect of statin treatment in pooled phase II and phase III baricitinib studies. Ann Rheum Dis. 2018 Jul;77(7):988-995. doi: 10.1136/annrheumdis-2017-212461. Epub 2018 Feb 20. PMID 29463520
- [Derived] Keystone EC, Genovese MC, Schlichting DE, de la Torre I, Beattie SD, Rooney TP, Taylor PC. Safety and Efficacy of Baricitinib Through 128 Weeks in an Open-label, Longterm Extension Study in Patients with Rheumatoid Arthritis. J Rheumatol. 2018 Jan;45(1):14-21. doi: 10.3899/jrheum.161161. Epub 2017 Aug 15. PMID 28811354
- [Derived] Keystone EC, Taylor PC, Drescher E, Schlichting DE, Beattie SD, Berclaz PY, Lee CH, Fidelus-Gort RK, Luchi ME, Rooney TP, Macias WL, Genovese MC. Safety and efficacy of baricitinib at 24 weeks in patients with rheumatoid arthritis who have had an inadequate response to methotrexate. Ann Rheum Dis. 2015 Feb;74(2):333-40. doi: 10.1136/annrheumdis-2014-206478. Epub 2014 Nov 27. PMID 25431052

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of 4 parts and a follow-up up to 28 days post the last dose of study drug.
Groups:
- 1 Milligrams (mg) LY3009104 QD - Part A: Administered orally once daily (QD) for 12 weeks in Part A.
  Methotrexate (MTX) was administered orally as background therapy.
- 2 mg LY3009104 QD - Parts A and B; 4 mg LY3009104 QD - Parts A and B; 8 mg LY3009104 QD - Parts A and B: Administered orally QD for 24 weeks in Parts A and B.
  MTX was administered orally as background therapy.
- Placebo QD - Part A: Placebo administered orally QD for 12 weeks in Part A.
  MTX was administered orally as background therapy.
- 2 mg LY3009104 BID - Part B: Participants who received Placebo or 1 mg LY3009104 in Part A were re-randomized at Week 12 to receive 2 mg LY3009104 twice daily (BID) in Part B.
  MTX was administered orally as background therapy.
- 4 mg LY3009104 QD - Part B: Participants who received Placebo or 1 mg LY3009104 in Part A were re-randomized at Week 12 to receive 4 mg LY3009104 QD in Part B.
  MTX was administered orally as background therapy.
- 4 mg LY3009104 QD - Parts C and D: Participants who received 2 mg LY3009104 QD or BID in Part B were re-assigned at Week 24 to 4 mg LY3009104 QD in Part C.
  Participants who received 4 mg LY3009104 QD in Part B continued to receive 4 mg LY3009104 QD in Part C.
  Participants who completed Part C continued to receive 4 mg LY3009104 QD in Part D.
  MTX was administered orally as background therapy.
- 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D: Participants who received 2 mg LY3009104 QD or BID in Part B were re-assigned at Week 24 to 4 mg LY3009104 QD in Part C.
  Participants who received 4 mg LY3009104 QD in Part B continued to receive 4 mg LY3009104 QD in Part C.
  At Weeks 28 and 32, participants who met dose escalation criteria received 8 mg LY3009104 QD for the rest of the Part C.
  Dose escalation criteria: ≥ 6 tender and 6 swollen joints based on the 28-joint count assessments and the clinical judgment of the investigator.
  Participants who completed Part C received 4 mg LY3009104 QD in Part D.
  MTX was administered orally as background therapy.
- 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D: Participants who received 8 mg LY3009104 QD in Part B remained on 8 mg LY3009104 QD in Part C.
  Participants who completed Part C received 4 mg LY3009104 QD in Part D.
  MTX was administered orally as background therapy.
Period: Part A (Weeks 0 Through 12)
Arm/Group | 1 Milligrams (mg) LY3009104 QD - Part A | 2 mg LY3009104 QD - Parts A and B | 4 mg LY3009104 QD - Parts A and B | 8 mg LY3009104 QD - Parts A and B | Placebo QD - Part A | 2 mg LY3009104 BID - Part B | 4 mg LY3009104 QD - Part B | 4 mg LY3009104 QD - Parts C and D | 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D | 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D
Started | 49 | 52 | 52 | 50 | 98 | 0 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 49 | 52 | 52 | 50 | 98 | 0 | 0 | 0 | 0 | 0
Completed | 44 | 51 | 50 | 49 | 82 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 1 | 2 | 1 | 16 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 1 | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Entry Criteria Not Met | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Period: Part B (Weeks 12 Through 24)
Arm/Group | 1 Milligrams (mg) LY3009104 QD - Part A | 2 mg LY3009104 QD - Parts A and B | 4 mg LY3009104 QD - Parts A and B | 8 mg LY3009104 QD - Parts A and B | Placebo QD - Part A | 2 mg LY3009104 BID - Part B | 4 mg LY3009104 QD - Part B | 4 mg LY3009104 QD - Parts C and D | 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D | 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D
Started | 0 | 51 | 50 | 49 | 0 | 63 | 63 | 0 | 0 | 0
Completed | 0 | 50 | 48 | 45 | 0 | 59 | 57 | 0 | 0 | 0
Not Completed | 0 | 1 | 2 | 4 | 0 | 4 | 6 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 0 | 3 | 4 | 0 | 0 | 0
Not completed — Entry Criteria Not Met | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Part C (Weeks 24 Through 76)
Arm/Group | 1 Milligrams (mg) LY3009104 QD - Part A | 2 mg LY3009104 QD - Parts A and B | 4 mg LY3009104 QD - Parts A and B | 8 mg LY3009104 QD - Parts A and B | Placebo QD - Part A | 2 mg LY3009104 BID - Part B | 4 mg LY3009104 QD - Part B | 4 mg LY3009104 QD - Parts C and D | 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D | 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 108 | 61 | 32
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 92 | 53 | 24
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 8 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Entry Criteria Not Met | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Reason missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Part D (Weeks 76 Through 128)
Arm/Group | 1 Milligrams (mg) LY3009104 QD - Part A | 2 mg LY3009104 QD - Parts A and B | 4 mg LY3009104 QD - Parts A and B | 8 mg LY3009104 QD - Parts A and B | Placebo QD - Part A | 2 mg LY3009104 BID - Part B | 4 mg LY3009104 QD - Part B | 4 mg LY3009104 QD - Parts C and D | 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D | 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 79 | 47 | 18
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 76 | 40 | 17
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- 1 mg LY3009104: Administered orally QD for initial 12 weeks (Part A) followed by randomization to either 4 mg QD or 2 mg BID for an additional 12 weeks (Part B). After 24 weeks of treatment, participants were eligible to participate in an open-label extension period (Part C). Part C: 4 mg or 8 mg administered orally QD for 52 weeks. After 76 weeks of treatment, participants were eligible to participate in an additional open-label extension period (Part D). Part D: 4 mg administered orally QD for 52 additional weeks.
  MTX was administered orally as background therapy.
- 2 mg LY3009104; 4 mg LY3009104: Administered orally QD for 24 weeks (Parts A and B). After 24 weeks of treatment, participants were eligible to participate in an open-label extension period (Part C). Part C: 4 mg or 8 mg administered orally QD for 52 weeks. After 76 weeks of treatment, participants were eligible to participate in an additional open-label extension period (Part D). Part D: 4 mg administered orally QD for 52 additional weeks.
  MTX was administered orally as background therapy.
- 8 mg LY3009104: Administered orally QD for 24 weeks (Parts A and B). After 24 weeks of treatment, participants were eligible to participate in an open-label extension period (Part C). Part C: 8 mg administered orally QD for 52 weeks. After 76 weeks of treatment, participants were eligible to participate in an additional open-label extension period (Part D). Part D: 4 mg administered orally QD for 52 additional weeks.
  MTX was administered orally as background therapy.
- Placebo: Placebo administered orally QD for initial 12 weeks (Part A) followed by randomization to either 4 mg QD or 2 mg BID for an additional 12 weeks (Part B). After 24 weeks of treatment, participants were eligible to participate in an open-label extension period (Part C). Part C: 4 mg or 8 mg administered orally QD for 52 weeks. After 76 weeks of treatment participants were eligible to participate in an additional open-label extension period (Part D). Part D: 4 mg administered orally QD for 52 additional weeks.
  MTX was administered orally as background therapy.
- Total: Total of all reporting groups
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo | Total
Number analyzed (Participants) | 49 | 52 | 52 | 50 | 98 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (11.07) | 50.7 (13.12) | 52.5 (10.42) | 52.7 (10.91) | 49.2 (12.15) | 51.2 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 44 | 37 | 41 | 85 | 249
  Male | 7 | 8 | 15 | 9 | 13 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 12 | 11 | 16 | 56
  Not Hispanic or Latino | 36 | 41 | 36 | 36 | 78 | 227
  Unknown or Not Reported | 3 | 4 | 4 | 3 | 4 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 3 | 2 | 7 | 19
  Asian | 8 | 8 | 7 | 9 | 15 | 47
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 2 | 6 | 11
  White | 37 | 40 | 40 | 37 | 70 | 224
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 16 | 16 | 31 | 95
  Hungary | 3 | 3 | 3 | 2 | 2 | 13
  Czech Republic | 4 | 3 | 6 | 3 | 7 | 23
  Mexico | 7 | 8 | 8 | 8 | 16 | 47
  Poland | 4 | 5 | 6 | 7 | 11 | 33
  Ukraine | 6 | 6 | 5 | 3 | 9 | 29
  Croatia | 0 | 1 | 0 | 1 | 5 | 7
  Romania | 2 | 2 | 1 | 3 | 3 | 11
  India | 7 | 8 | 7 | 7 | 14 | 43
Duration of Rheumatoid Arthritis [Mean (Standard Deviation); unit: years] | 5.45 (3.885) | 5.53 (4.377) | 5.28 (4.466) | 6.63 (5.048) | 5.40 (4.283) | 5.62 (4.401)
Tender Joint Counts (TJC) [Mean (Standard Deviation); unit: number of joints] — TJC is the number of tender and painful joints determined for each participant by examination of 68 joints. Joints were assessed by pressure and joint manipulation on physical examination. Participants were asked for pain sensations on these manipulations and watched for spontaneous pain reactions. Any positive response on pressure, movement, or both was translated into a single tender-versus-nontender dichotomy.
  number of joints | 21.4 (10.90) | 23.0 (12.60) | 19.9 (12.71) | 24.4 (13.76) | 22.2 (12.06) | 22.2 (12.38)
Swollen Joint Counts (SJC) [Mean (Standard Deviation); unit: number of joints] — SJC is the number of swollen joints determined for each participant by examination of 66 joints. Joints were classified as either swollen or not swollen. Swelling was defined as palpable fluctuating synovitis of the joint.
  number of joints | 15.2 (6.55) | 17.0 (9.32) | 14.8 (7.54) | 16.1 (7.92) | 15.8 (8.64) | 15.8 (8.13)
High Sensitivity C-Reactive Protein (hsCRP) [Mean (Standard Deviation); unit: milligrams/liter (mg/L)] — HsCRP is a laboratory analyte that is an indicator of inflammation. Decreases in hsCRP represent reductions in inflammation. Population: All randomized participants who received at least one dose of study drug and had evaluable hsCRP data at baseline.
  milligrams/liter (mg/L)
    number analyzed (Participants) | 49 | 52 | 52 | 50 | 97 | 300
    (all) | 11.22 (12.410) | 12.02 (22.111) | 11.39 (16.941) | 14.32 (15.602) | 14.03 (23.527) | 12.81 (19.402)
Erythrocyte Sedimentation Rate (ESR) [Mean (Standard Deviation); unit: millimeters/hour (mm/hr)] — ESR is a laboratory analyte that is an indicator of inflammation. Decreases represent reductions in inflammation.
  millimeters/hour (mm/hr) | 38.2 (17.57) | 36.5 (14.62) | 35.4 (17.16) | 43.3 (18.17) | 39.9 (20.94) | 38.8 (18.39)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in the 4 mg and 8 mg Dose Groups Who Achieved an American College of Rheumatology 20 (ACR20) Responder Index Response Baseline Through Week 12
Description: ACR20 Responder Index is a composite of clinical, laboratory, and functional measures in rheumatoid arthritis (RA). An ACR20 Responder is a participant who had ≥20% improvement from baseline in both 68 tender and 66 swollen joint counts and ≥20% improvement in at least 3 of 5 criteria: Patient's and Physician's Global Assessment of Disease Activity, Health Assessment Questionnaire-Disability Index (HAQ-DI) (assessment of participant's physical function), pain due to RA, and hsCRP. Participants who discontinue before analysis time point are treated as non-responders. Percentage of participants achieving ACR20 response = (number of ACR20 responders) / (number of participants analyzed) * 100.
Time Frame: Baseline through Week 12
Population: All randomized participants who received placebo, 4 mg or 8 mg LY3009104 in Part A. Participants who had missing components of the ACR20 index at Week 12 had these components imputed by last observation carried forward (LOCF).
Measure: Number; unit: percentage of participants
Groups:
- 4 or 8 mg LY3009104: 4 or 8 mg LY3009104 administered orally QD for 12 weeks in Part A.
  MTX was administered orally as background therapy.
- Placebo: Placebo administered orally QD for 12 weeks in Part A.
  MTX was administered orally as background therapy.
Arm/Group | 4 or 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 102 | 98
percentage of participants | 76 | 41
Statistical Analysis 1: Comparison: 4 or 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — A priori p-value significance threshold: 1-sided ≤0.10

2. Secondary Outcome: Percentage of Participants Who Achieved an ACR20 Responder Index Response Baseline Through Week 12 - Model Based Dose Response
Description: ACR20 Responder Index is a composite of clinical, laboratory, and functional measures in RA. An ACR20 Responder is a participant who had ≥20% improvement from baseline in both 68 tender and 66 swollen joint counts and ≥20% improvement in at least 3 of 5 criteria: Patient's and Physician's Global Assessment of Disease Activity, HAQ-DI (assessment of participant's physical function), pain due to RA, and hsCRP. Participants who discontinue before analysis time point are treated as non-responders. Percentage of participants achieving ACR20 response = (number of ACR20 responders) / (number of participants analyzed) * 100. Data presented are model-based Bayesian posterior mean response rates with 95% credible interval.
Time Frame: Baseline through Week 12
Population: All randomized participants who received study drug in Part A. Participants who had missing components of the ACR20 index at Week 12 had these components imputed by LOCF.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 1 mg LY3009104: 1 mg LY3009104 administered orally QD for 12 weeks in Part A.
  MTX was administered orally as background therapy.
- 2 mg LY3009104: 2 mg LY3009104 administered orally QD for 12 weeks in Part A.
  MTX was administered orally as background therapy.
- 4 mg LY3009104: 4 mg LY3009104 administered orally QD for 12 weeks in Part A.
  MTX was administered orally as background therapy.
- 8 mg LY3009104: 8 mg LY3009104 administered orally QD for 12 weeks in Part A.
  MTX was administered orally as background therapy.
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 49 | 52 | 52 | 50 | 98
percentage of participants | 54.6 [42.2 to 67.1] | 55.2 [42.3 to 67.6] | 74.3 [63.1 to 84.1] | 77.2 [65.9 to 86.7] | 42.1 [32.9 to 51.6]

3. Secondary Outcome: Percentage of Participants Who Achieved an ACR20 Responder Index Response Baseline Through Week 24
Description: ACR20 Responder Index is a composite of clinical, laboratory, and functional measures in RA. An ACR20 Responder is a participant who had ≥20% improvement from baseline in both 68 tender and 66 swollen joint counts and ≥20% improvement in at least 3 of 5 criteria: Patient's and Physician's Global Assessment of Disease Activity, HAQ-DI (assessment of participant's physical function), pain due to RA, and hsCRP. Participants who discontinue before analysis time points are treated as non-responders. Percentage of participants achieving ACR20 response = (number of ACR20 responders) / (number of participants treated) * 100.
Time Frame: Baseline through Weeks 2, 4, 8, 12, 16, 20, 24
Population: All randomized participants who received study drug in Parts A and B. Participants who had missing components of the ACR20 index at analysis time points had these components imputed by LOCF.
Measure: Number; unit: percentage of participants
Groups:
- 2 mg LY3009104: 2 mg LY3009104 administered orally QD for 24 weeks in Parts A and B.
  MTX was administered orally as background therapy.
- 4 mg LY3009104: 4 mg LY3009104 administered orally QD for 24 weeks in Parts A and B.
  MTX was administered orally as background therapy.
- 8 mg LY3009104: 8 mg LY3009104 administered orally QD for 24 weeks in Parts A and B.
  MTX was administered orally as background therapy.
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 49 | 52 | 52 | 50 | 98
percentage of participants
  Week 2 | 29 | 21 | 42 | 44 | 11
  Week 4 | 43 | 37 | 60 | 54 | 24
  Week 8 | 43 | 42 | 67 | 72 | 36
  Week 12 | 57 | 54 | 75 | 78 | 41
  Week 16 | NA — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore percentage was not calculated. | 63 | 67 | 64 | NA — Participants were not dosed with placebo after Week 12, therefore percentage was not calculated.
  Week 20 | NA — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore percentage was not calculated. | 71 | 77 | 78 | NA — Participants were not dosed with placebo after Week 12, therefore percentage was not calculated.
  Week 24 | NA — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore percentage was not calculated. | 62 | 75 | 72 | NA — Participants were not dosed with placebo after Week 12, therefore percentage was not calculated.
Statistical Analysis 1: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.045, Fisher Exact — P-value is for Week 12. A priori p-value significance threshold: 1-sided ≤0.10
Statistical Analysis 2: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.088, Fisher Exact — P-value is for Week 12. A priori p-value significance threshold: 1-sided ≤0.10
Statistical Analysis 3: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact — P-value is for Week 12. A priori p-value significance threshold: 1-sided ≤0.10
Statistical Analysis 4: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact — P-value is for Week 12. A priori p-value significance threshold: 1-sided ≤0.10

4. Secondary Outcome: Percentage of Participants Who Achieved an ACR20 Response Baseline Through Weeks 76 and 128
Description: ACR20 Responder Index is a composite of clinical, laboratory, and functional measures in RA. An ACR20 Responder is a participant who had ≥20% improvement from baseline in both 68 tender and 66 swollen joint counts and ≥20% improvement in at least 3 of 5 criteria: Patient's and Physician's Global Assessment of Disease Activity, HAQ-DI (assessment of participant's physical function), pain due to RA, and hsCRP. Participants who discontinue before analysis time points are treated as non-responders. Percentage of participants achieving ACR20 response = (number of ACR20 responders) / (number of participants analyzed) * 100.
Time Frame: Baseline through Weeks 76 and 128
Population: All participants who received study drug in Parts C and D. Participants who had missing components of the ACR20 index at analysis time points had these components imputed by LOCF.
Measure: Number; unit: percentage of participants
Groups:
- 4 mg LY3009104 QD - Parts C and D: Received Placebo, or 1 mg, or 2 mg, or 4 mg LY3009104 in Part A.
  Received 2 mg LY3009104 QD, or BID, or 4 mg LY3009104 QD in Part B.
  Received 4 mg LY3009104 QD in Part C.
  Received 4 mg LY3009104 QD in Part D.
  MTX was administered orally as background therapy.
- 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D: Received Placebo, or 1 mg, or 2 mg, or 4 mg LY3009104 in Part A.
  Received 2 mg LY3009104 QD, or BID, or 4 mg LY3009104 QD in Part B.
  Received 4 mg LY3009104 QD in Part C. During Part C, at Weeks 28 and 32, participants who met dose escalation criteria received 8 mg LY3009104 QD for the rest of the Part C.
  Dose escalation criteria: ≥6 tender and 6 swollen joints based on the 28-joint count assessments and the clinical judgment of the investigator.
  Received 4 mg LY3009104 QD in Part D.
  MTX was administered orally as background therapy.
- 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D: Received 8 mg LY3009104 QD in Parts A, B and C.
  Received 4 mg LY3009104 QD in Part D.
  MTX was administered orally as background therapy.
Arm/Group | 4 mg LY3009104 QD - Parts C and D | 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D | 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D
Number analyzed (Participants) | 108 | 61 | 32
percentage of participants
  Week 76 (n=108, 61, 32) | 71 | 67 | 59
  Week 128 (n=79, 47, 18) | 77 | 57 | 72

5. Secondary Outcome: Percentage of Participants Who Achieved an ACR 50 Responder Index Response Baseline Through Week 24
Description: ACR50 Responder Index is a composite of clinical, laboratory, and functional measures in RA. An ACR50 Responder is a participant who had ≥50% improvement from baseline in both 68 tender and 66 swollen joint counts and ≥50% improvement in at least 3 of 5 criteria: Patient's and Physician's Global Assessment of Disease Activity, HAQ-DI (assessment of participant's physical function), pain due to RA, and hsCRP. Participants who discontinue before analysis time points are treated as non-responders. Percentage of participants achieving ACR50 response = (number of ACR50 responders) / (number of participants analyzed) * 100.
Time Frame: Baseline through Weeks 2, 4, 8, 12, 16, 20, 24
Population: All randomized participants who received study drug in Parts A and B. Participants who had missing components of the ACR50 index at analysis time points had these components imputed by LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 49 | 52 | 52 | 50 | 98
percentage of participants
  Week 2 | 0 | 4 | 21 | 4 | 2
  Week 4 | 10 | 10 | 29 | 22 | 3
  Week 8 | 16 | 10 | 33 | 36 | 7
  Week 12 | 31 | 17 | 35 | 40 | 10
  Week 16 | NA — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore percentage was not calculated. | 19 | 38 | 44 | NA — Participants were not dosed with placebo after Week 12, therefore percentage was not calculated.
  Week 20 | NA — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore percentage was not calculated. | 27 | 46 | 48 | NA — Participants were not dosed with placebo after Week 12, therefore percentage was not calculated.
  Week 24 | NA — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore percentage was not calculated. | 19 | 46 | 54 | NA — Participants were not dosed with placebo after Week 12, therefore percentage was not calculated.
Statistical Analysis 1: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.003, Fisher Exact — P-value is for Week 12. A priori p-value significance threshold: 1-sided ≤0.10
Statistical Analysis 2: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.162, Fisher Exact — P-value is for Week 12. A priori p-value significance threshold: 1-sided ≤0.10
Statistical Analysis 3: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact — P-value is for Week 12. A priori p-value significance threshold: 1-sided ≤0.10
Statistical Analysis 4: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact — P-value is for Week 12. A priori p-value significance threshold: 1-sided ≤0.10

6. Secondary Outcome: Percentage of Participants Who Achieved an ACR50 Response Baseline Through Weeks 76 and 128
Description: as for outcome 5
Time Frame: Baseline through Weeks 76 and 128
Population: All participants who received study drug in Parts C and D. Participants who had missing components of the ACR50 index at analysis time points had these components imputed by LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | 4 mg LY3009104 QD - Parts C and D | 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D | 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D
Number analyzed (Participants) | 108 | 61 | 32
percentage of participants
  Week 76 (n=108, 61, 32) | 49 | 41 | 44
  Week 128 (n=79, 47, 18) | 58 | 30 | 44

7. Secondary Outcome: Percentage of Participants Who Achieved an ACR70 Responder Index Response Baseline Through Week 24
Description: ACR70 Responder Index is a composite of clinical, laboratory, and functional measures in RA. An ACR70 Responder is a participant who had ≥70% improvement from baseline in both 68 tender and 66 swollen joint counts and ≥70% improvement in at least 3 of 5 criteria: Patient's and Physician's Global Assessment of Disease Activity, HAQ-DI (assessment of participant's physical function), pain due to RA, and hsCRP. Participants who discontinue before analysis time points are treated as non-responders. Percentage of participants achieving ACR70 response = (number of ACR70 responders) / (number of participants analyzed) * 100.
Time Frame: Baseline through Weeks 2, 4, 8, 12, 16, 20, 24
Population: All randomized participants who received study drug in Parts A and B. Participants who had missing components of the ACR70 index at analysis time points had these components imputed by LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 49 | 52 | 52 | 50 | 98
percentage of participants
  Week 2 | 0 | 2 | 12 | 0 | 0
  Week 4 | 2 | 4 | 10 | 6 | 0
  Week 8 | 4 | 4 | 15 | 22 | 0
  Week 12 | 12 | 8 | 23 | 20 | 2
  Week 16 | NA — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore percentage was not calculated. | 8 | 23 | 30 | NA — Participants were not dosed with placebo after Week 12, therefore percentage was not calculated.
  Week 20 | NA — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore percentage was not calculated. | 10 | 21 | 26 | NA — Participants were not dosed with placebo after Week 12, therefore percentage was not calculated.
  Week 24 | NA — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore percentage was not calculated. | 10 | 27 | 24 | NA — Participants were not dosed with placebo after Week 12, therefore percentage was not calculated.
Statistical Analysis 1: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.017, Fisher Exact — P-value is for Week 12. A priori p-value significance threshold: 1-sided ≤0.10
Statistical Analysis 2: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.109, Fisher Exact — P-value is for Week 12. A priori p-value significance threshold: 1-sided ≤0.10
Statistical Analysis 3: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact — P-value is for Week 12. A priori p-value significance threshold: 1-sided ≤0.10
Statistical Analysis 4: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact — P-value is for Week 12. A priori p-value significance threshold: 1-sided ≤0.10

8. Secondary Outcome: Percentage of Participants Who Achieved an ACR70 Response Baseline Through Weeks 76 and 128
Description: as for outcome 7
Time Frame: Baseline through Weeks 76 and 128
Population: All participants who received study drug in Parts C and D. Participants who had missing components of the ACR70 index at analysis time points had these components imputed by LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | 4 mg LY3009104 QD - Parts C and D | 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D | 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D
Number analyzed (Participants) | 108 | 61 | 32
percentage of participants
  Week 76 (n=108, 61, 32) | 29 | 18 | 25
  Week 128 (n=79, 47, 18) | 28 | 17 | 22

9. Secondary Outcome: Percentage of Participants Who Achieved an ACR50 Response Baseline Through Week 12 - Model Based Dose Response
Description: ACR50 Responder Index is a composite of clinical, laboratory, and functional measures in RA. An ACR50 Responder is a participant who had ≥50% improvement from baseline in both 68 tender and 66 swollen joint counts and ≥50% improvement in at least 3 of 5 criteria: Patient's and Physician's Global Assessment of Disease Activity, HAQ-DI (assessment of participant's physical function), pain due to RA, and hsCRP. Participants who discontinue before analysis time point are treated as non-responders. Percentage of participants achieving ACR50 response = (number of ACR50 responders) / (number of participants analyzed) * 100. Data presented are model-based Bayesian posterior mean response rates with 95% credible interval.
Time Frame: Baseline through Week 12
Population: All randomized participants who received study drug in Part A. Participants who had missing components of the ACR50 index at analysis time point had these components imputed by LOCF.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 49 | 52 | 52 | 50 | 98
percentage of participants | 26.5 [16.0 to 39.2] | 18.8 [9.9 to 29.7] | 34.4 [23.1 to 46.7] | 39.2 [27.1 to 52.2] | 12.0 [6.5 to 18.8]

10. Secondary Outcome: ACR Percent Improvement (ACR-N)
Description: ACR-N is a continuous measure of clinical, laboratory, and functional outcomes in RA that characterizes percentage (%) of improvement in disease activity from baseline based on ACR core set. This index was calculated as minimum of a) % of improvement in TJC, b) % of improvement in SJC, and c) third highest percentage of improvement of remaining 5 ACR core criteria: If ≥3 components of the 5 ACR core criteria were missing, then c) was set to missing; if any of 3 components a), b), or c) were missing, then ACR-N was set to missing. Percentage of improvement was truncated to a range of -100 to 100 to minimize impact of outliers (greater scores indicate greater % improvement) and negative scores indicate a decline. Data presented are model-based Bayesian posterior mean response rates with 95% credible interval.
Time Frame: Baseline through Week 12
Population: All randomized participants who received study drug in Part A. Participants who had missing components of the ACR-N at Week 12 had these components imputed by LOCF.
Measure: Number (95% Confidence Interval); unit: percentage of improvement
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 49 | 52 | 52 | 50 | 98
percentage of improvement | 17.30 [7.57 to 28.22] | 19.42 [8.74 to 29.25] | 28.59 [17.67 to 40.83] | 29.00 [17.67 to 41.47] | 10.97 [-0.39 to 21.64]

11. Secondary Outcome: Mean Change From Baseline to Weeks 12 and 24 in Tender and Swollen Joint Counts (TJC and SJC)
Description: TJC is the number of tender and painful joints determined for each participant by examination of 68 joints. Joints were assessed by pressure and joint manipulation on physical examination. Participants were asked for pain sensations on these manipulations and watched for spontaneous pain reactions. Any positive response on pressure, movement, or both was translated into a single tender-versus-nontender dichotomy. SJC is the number of swollen joints determined for each participant by examination of 66 joints. Joints were classified as either swollen or not swollen. Swelling was defined as palpable fluctuating synovitis of the joint.
Time Frame: Baseline, Weeks 12 and 24
Population: All randomized participants who received study drug in Parts A and B and had TJC and SJC evaluated at analysis time points. LOCF was used to impute missing post-baseline values
Measure: Mean (Standard Deviation); unit: number of joints
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 49 | 52 | 51 | 50 | 98
number of joints
  TJC - Week 12 | -8.4 (12.70) | -11.3 (13.50) | -12.2 (10.45) | -14.7 (12.97) | -7.6 (12.31)
  TJC - Week 24 | NA (NA) — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore mean and standard deviation (SD) were not calculated. | -12.4 (12.60) | -14.0 (9.54) | -17.5 (11.23) | NA (NA) — Participants were not dosed with placebo after Week 12, therefore mean and SD were not calculated.
  SJC - Week 12 | -8.1 (7.24) | -8.9 (9.03) | -9.6 (6.49) | -10.4 (8.88) | -6.7 (7.97)
  SJC - Week 24 | NA (NA) — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore mean and SD were not calculated. | -10.0 (8.16) | -10.5 (6.42) | -12.2 (7.29) | NA (NA) — Participants were not dosed with placebo after Week 12, therefore mean and SD were not calculated.
Statistical Analysis 1: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.480, ANCOVA — P-value is for TJC - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 2: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.064, ANCOVA — P-value is for TJC - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 3: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for TJC - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 4: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value is for TJC - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 5: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.116, ANCOVA — P-value is for SJC - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 6: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.201, ANCOVA — P-value is for SJC - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 7: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for SJC - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 8: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value is for SJC - Week 12. A priori p-value significance threshold: 2-sided ≤0.10

12. Secondary Outcome: Mean Change From Baseline to Weeks 76 and 128 in TJC and SJC
Description: as for outcome 11
Time Frame: Baseline, Weeks 76 and 128
Population: All participants who received study drug in Parts C and D and had TJC and SJC evaluated at analysis time points. LOCF was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 4 mg LY3009104 QD - Parts C and D | 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D | 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D
Number analyzed (Participants) | 108 | 61 | 32
units on a scale
  TJC - Week 76 (n=108, 61, 32) | -15.7 (11.26) | -16.0 (13.37) | -18.1 (12.06)
  TJC - Week 128 (n=79, 47, 18) | -16.4 (11.01) | -15.3 (12.56) | -14.0 (13.68)
  SJC - Week 76 (n=108, 61, 32) | -11.6 (6.40) | -12.9 (7.80) | -12.4 (7.67)
  SJC - Week 128 (n=79, 47, 18) | -11.4 (6.81) | -12.4 (8.01) | -11.6 (6.23)

13. Secondary Outcome: Mean Change From Baseline to Weeks 12 and 24 in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: The HAQ-DI questionnaire assesses the participant's self-perception on the degree of difficulty [0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do)] when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area were averaged to calculate HAQ-DI scores, which ranged from 0 (no disability) to 3 (worst disability). A decrease in HAQ-DI score indicated an improvement in the participant's condition.
Time Frame: Baseline, Weeks 12 and 24
Population: All randomized participants who received study drug in Parts A and B and had HAQ-DI evaluated at analysis time points. LOCF was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 49 | 52 | 51 | 50 | 98
units on a scale
  Week 12 | -0.35 (0.528) | -0.18 (0.524) | -0.33 (0.459) | -0.39 (0.497) | -0.10 (0.406)
  Week 24 | NA (NA) — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore mean and SD were not calculated. | -0.18 (0.505) | -0.32 (0.506) | -0.44 (0.529) | NA (NA) — Participants were not dosed with placebo after Week 12, therefore mean and SD were not calculated.
Statistical Analysis 1: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 2: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.167, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 3: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 4: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10

14. Secondary Outcome: Mean Change From Baseline to Weeks 76 and 128 in HAQ-DI Score
Description: as for outcome 13
Time Frame: Baseline, Weeks 76 and 128
Population: All participants who received study drug in Parts C and D and had HAQ-DI evaluated at analysis time points. LOCF was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 4 mg LY3009104 QD - Parts C and D | 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D | 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D
Number analyzed (Participants) | 108 | 61 | 32
units on a scale
  Week 76 (n=108, 61, 32) | -0.34 (0.58) | -0.29 (0.53) | -0.55 (0.58)
  Week 128 (n=79, 47, 18) | -0.31 (0.61) | -0.22 (0.56) | -0.30 (0.66)

15. Secondary Outcome: Mean Change From Baseline to Weeks 12 and 24 in High-Sensitivity C-Reactive Protein (hsCRP)
Description: hsCRP is a laboratory analyte that is an indicator of inflammation. Decreases in hsCRP represent reductions in inflammation.
Time Frame: Baseline, Weeks 12 and 24
Population: All randomized participants who received study drug in Parts A and B and had hsCRP evaluated at analysis time points. LOCF was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 49 | 52 | 51 | 50 | 97
mg/L
  Week 12 | -6.14 (10.236) | -3.39 (19.409) | -7.06 (16.945) | -2.32 (32.582) | 1.50 (34.107)
  Week 24 | NA (NA) — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore mean and SD were not calculated. | -4.76 (18.695) | -4.95 (19.819) | -7.61 (17.548) | NA (NA) — Participants were not dosed with placebo after Week 12, therefore mean and SD were not calculated.
Statistical Analysis 1: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.016, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 2: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.108, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 3: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.008, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 4: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.368, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10

16. Secondary Outcome: Mean Change From Baseline to Weeks 76 and 128 in hsCRP
Description: as for outcome 15
Time Frame: Baseline, Weeks 76 and 128
Population: All participants who received study drug in Parts C and D and had hsCRP evaluated at analysis time points. LOCF was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 4 mg LY3009104 QD - Parts C and D | 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D | 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D
Number analyzed (Participants) | 108 | 61 | 32
mg/L
  Week 76 (n=108, 61, 32) | -3.9 (22.43) | -3.3 (14.28) | -2.9 (25.36)
  Week 128 (n=79, 47, 18) | -6.8 (13.66) | -2.9 (21.88) | -8.2 (12.33)

17. Secondary Outcome: Mean Change From Baseline to Weeks 12 and 24 in Erythrocyte Sedimentation Rate (ESR)
Description: ESR is a laboratory analyte that is an indicator of inflammation. Decreases represent reductions in inflammation.
Time Frame: Baseline, Weeks 12 and 24
Population: All randomized participants who received study drug in Parts A and B and had ESR evaluated at analysis time points.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 44 | 51 | 50 | 49 | 83
mm/hr
  Week 12 (n=44, 51, 50, 49, 83) | -11.6 (14.45) | -6.4 (16.81) | -11.5 (17.28) | -13.9 (22.42) | -6.0 (19.49)
  Week 24 (n=0, 50, 48, 45, 0) | NA (NA) — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore mean and SD were not calculated. | -6.9 (13.89) | -9.2 (19.00) | -13.7 (21.62) | NA (NA) — Participants were not dosed with placebo after Week 12, therefore mean and SD were not calculated.
Statistical Analysis 1: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.039, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 2: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.458, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 3: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.008, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 4: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.029, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10

18. Secondary Outcome: Mean Change From Baseline to Weeks 76 and 128 in ESR
Description: ESR is a laboratory analyte that is an indicator of inflammation. Decreases represent reductions in inflammation.
Time Frame: Baseline, Weeks 76 and 128
Population: All participants who received study drug in Parts C and D and had ESR evaluated at analysis time points. LOCF was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | 4 mg LY3009104 QD - Parts C and D | 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D | 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D
Number analyzed (Participants) | 108 | 61 | 32
mm/hr
  Week 76 (n=108, 61, 32) | -13.0 (18.84) | -7.4 (26.28) | -8.9 (23.12)
  Week 128 (n=79, 47, 18) | -16.0 (18.74) | -8.5 (23.11) | -15.5 (23.07)

19. Secondary Outcome: Mean Change From Baseline to Weeks 12 and 24 in Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity and Patient's Assessment of Pain
Description: Physician's and Patient's Assessments of Disease Activity (DA) assessed using a visual analog scale (VAS) that ranged from 0 to 100 millimeters (mm), where 0 indicated no arthritis activity and 100 indicated extremely active arthritis. Patient's assessment of pain due to arthritis was also assessed using a VAS that ranged from 0 (no pain) to 100 mm (worst possible pain).
Time Frame: Baseline, Weeks 12 and 24
Population: All randomized participants who received study drug in Parts A and B and had physician's and participant's assessments of disease activity and participant's pain evaluated at analysis time points. LOCF was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 49 | 52 | 51 | 50 | 98
units on a scale
  Physician's Assessment of DA - Week 12 | -23.9 (18.49) | -25.0 (20.81) | -30.4 (18.75) | -33.5 (19.49) | -19.0 (21.40)
  Physician's Assessment of DA - Week 24 | NA (NA) — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore mean and SD were not calculated. | -27.8 (21.13) | -35.5 (17.72) | -37.8 (18.73) | NA (NA) — Participants were not dosed with placebo after Week 12, therefore mean and SD were not calculated.
  Patient's Assessment of DA - Week 12 | -24.9 (27.26) | -16.2 (22.43) | -25.4 (21.61) | -29.8 (21.20) | -10.3 (22.02)
  Patient's Assessment of DA - Week 24 | NA (NA) — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore mean and SD were not calculated. | -16.9 (24.96) | -30.2 (21.85) | -30.0 (20.90) | NA (NA) — Participants were not dosed with placebo after Week 12, therefore mean and SD were not calculated.
  Patient's Assessment of Pain - Week 12 | -22.8 (27.39) | -14.2 (17.82) | -25.0 (19.22) | -25.3 (20.31) | -8.8 (22.77)
  Patient's Assessment of Pain - Week 24 | NA (NA) — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore mean and SD were not calculated. | -14.7 (20.57) | -27.3 (22.11) | -26.9 (19.22) | NA (NA) — Participants were not dosed with placebo after Week 12, therefore mean and SD were not calculated.
Statistical Analysis 1: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.217, ANCOVA — P-value is for Physician's Assessment of DA - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 2: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.092, ANCOVA — P-value is for Physician's Assessment of DA - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 3: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Physician's Assessment of DA - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 4: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Physician's Assessment of DA - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 5: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Patient's Assessment of DA - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 6: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.072, ANCOVA — P-value is for Patient's Assessment of DA - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 7: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Patient's Assessment of DA - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 8: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Patient's Assessment of DA - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 9: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Patient's Assessment of Pain - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 10: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.082, ANCOVA — P-value is for Patient's Assessment of Pain - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 11: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Patient's Assessment of Pain - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 12: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Patient's Assessment of Pain - Week 12. A priori p-value significance threshold: 2-sided ≤0.10

20. Secondary Outcome: Mean Change From Baseline to Weeks 76 and 128 in Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity and Patient's Assessment of Pain
Description: Physician's and Patient's assessments of DA assessed using a VAS that ranged from 0 to 100 mm, where 0 indicated no arthritis activity and 100 indicated extremely active arthritis. Patient's assessment of pain due to arthritis assessed using a VAS that ranged from 0 (no pain) to 100 mm (worst possible pain).
Time Frame: Baseline, Weeks 76 and 128
Population: All participants who received study drug in Parts C and D and had physician's and participant's assessments of disease activity and pain evaluated at analysis time points. LOCF was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 4 mg LY3009104 QD - Parts C and D | 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D | 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D
Number analyzed (Participants) | 108 | 61 | 32
units on a scale
  Physician Assessment of DA-Week 76 (n=108, 61, 32) | -40.3 (19.15) | -32.3 (23.37) | -40.5 (21.44)
  Physician Assessment of DA-Week 128 (n=79, 47, 18) | -39.5 (20.32) | -31.0 (25.54) | -34.0 (27.51)
  Patient Assessment of DA-Week 76 (n=108, 61, 32) | -27.5 (26.49) | -27.5 (25.52) | -27.6 (24.11)
  Patient Assessment of DA-Week 128 (n=79, 47, 18) | -27.9 (27.40) | -19.3 (29.72) | -27.6 (25.17)
  Patient Assessment of Pain-Week 76 (n=108, 61, 32) | -25.1 (24.10) | -27.3 (24.24) | -23.4 (23.49)
  Patient Assessment of Pain-Week 128 (n=79, 47, 18) | -24.2 (24.35) | -18.0 (28.85) | -22.3 (22.99)

21. Secondary Outcome: Mean Change From Baseline to Weeks 12 and 24 in Disease Activity Score (DAS) Based on the 28 Diarthrodial Joint Count and CRP Level (DAS28-CRP)
Description: Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consisted of composite score of following variables: tender joint count-28 (TJC28), swollen joint count-28 (SJC28), CRP (mg/L), and Patient's Global Assessment of Disease Activity using VAS (patient's global VAS). DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*patient's global VAS+0.96. Scores ranged from 1.0-9.4, where lower scores indicated less disease activity, and remission was DAS28-CRP <2.6. A decrease in DAS28-CRP indicated an improvement in participant's condition.
Time Frame: Baseline, Weeks 12 and 24
Population: All randomized participants who received study drug in Parts A and B and had DAS28-CRP evaluated at analysis time points. LOCF was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 49 | 52 | 50 | 50 | 93
units on a scale
  Week 12 | -1.47 (1.299) | -1.40 (1.210) | -2.09 (1.220) | -2.15 (1.273) | -0.98 (1.141)
  Week 24 | NA (NA) — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore mean and SD were not calculated. | -1.53 (1.187) | -2.25 (1.054) | -2.47 (1.280) | NA (NA) — Participants were not dosed with placebo after Week 12, therefore mean and SD were not calculated.
Statistical Analysis 1: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.024, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 2: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.030, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 3: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 4: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10

22. Secondary Outcome: Mean Change From Baseline to Weeks 76 and 128 in DAS28-CRP
Description: Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), CRP (mg/L), and Patient's Global Assessment of Disease Activity using visual analog scale (VAS) (patient's global VAS). DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*patient's global VAS+0.96. Scores ranged from 1.0-9.4, where lower scores indicated less disease activity and remission is DAS28-CRP <2.6. A decrease in DAS28-CRP indicated an improvement in participant's condition.
Time Frame: Baseline, Weeks 76 and 128
Population: All participants who received study drug in Parts C and D and had DAS28-CRP evaluated at analysis time points. LOCF was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 4 mg LY3009104 QD - Parts C and D | 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D | 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D
Number analyzed (Participants) | 107 | 61 | 31
units on a scale
  Week 76 (n=107, 61, 31) | -2.47 (1.23) | -2.16 (1.28) | -2.68 (1.12)
  Week 128 (n=79, 47, 18) | -2.56 (1.16) | -2.02 (1.23) | -2.35 (1.40)

23. Secondary Outcome: Percentage of Responders According to European League Against Rheumatism Responder Index Based on 28-joint Count (EULAR28) Baseline Through Weeks 12 and 24
Description: EULAR28 categorizes clinical response based upon improvement since baseline in DAS modified to include the 28-joint count (DAS28) and post-baseline DAS28. DAS28 consists of a composite score of the following variables: TJC28, SJC28, CRP, and Patient's Global Assessment of their Disease Activity (patient's global VAS). DAS28 scores range from 1.0-9.4. EULAR28 categories include: No Response (improvement in DAS28 of ≤0.6 units or post-baseline DAS28 score >5.1 with improvement by ≤1.2 units), Moderate Response (post-baseline DAS28 ≤5.1 with improvement by >0.6 units but ≤1.2 units or post-baseline DAS28 score >3.2 with improvement by >1.2 units), and Good Response (post-baseline DAS28 score ≤3.2 with improvement by >1.2 units).
Time Frame: Baseline through Weeks 12 and 24
Population: All randomized participants who received study drug in Parts A and B and had EULAR28 evaluated at analysis time points.
Measure: Number; unit: percentage of participants
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 49 | 52 | 52 | 50 | 98
percentage of participants
  Good Response - Week 12 | 22 | 17 | 46 | 40 | 16
  Moderate Response - Week 12 | 43 | 63 | 31 | 46 | 35
  No Response - Week 12 | 35 | 19 | 23 | 14 | 49
  Good Response - Week 24 | NA — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore percentage was not calculated. | 25 | 42 | 46 | NA — Participants were not dosed with placebo after Week 12, therefore percentage was not calculated.
  Moderate Response - Week 24 | NA — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore percentage was not calculated. | 52 | 42 | 32 | NA — Participants were not dosed with placebo after Week 12, therefore percentage was not calculated.
  No Response - Week 24 | NA — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore percentage was not calculated. | 23 | 15 | 22 | NA — Participants were not dosed with placebo after Week 12, therefore percentage was not calculated.
Statistical Analysis 1: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.120, Cochran-Mantel-Haenszel — P-value is for comparison of the superiority of the LY3009104 dose level vs. placebo for the ordinal levels of response - Week 12. A priori p-value significance threshold: 1-sided ≤0.10
Statistical Analysis 2: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.012, Cochran-Mantel-Haenszel — [p-value comment as in outcome 23, analysis 1]
Statistical Analysis 3: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 23, analysis 1]
Statistical Analysis 4: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 23, analysis 1]

24. Secondary Outcome: Percentage of Responders According to EULAR28 Baseline Through Weeks 76 and 128
Description: EULAR28 categorizes clinical response based upon improvement since baseline in Disease Activity Score modified to include the 28-joint count (DAS28) and post-baseline DAS28. DAS28 consists of a composite score of the following variables: tender joint count (TJC28), swollen joint count (SJC28), CRP, and Patient's Global Assessment of their Disease Activity (patient's global VAS). DAS28 scores range from 1.0-9.4. EULAR28 categories include: No Response (improvement in DAS28 of ≤0.6 units or post-baseline DAS28 score >5.1 with improvement by ≤1.2 units), Moderate Response (post-baseline DAS28 ≤5.1 with improvement by >0.6 units but ≤1.2 units or post-baseline DAS28 score >3.2 with improvement by >1.2 units), and Good Response (post-baseline DAS28 score ≤3.2 with improvement by >1.2 units).
Time Frame: Baseline, Weeks 76 and 128
Population: All participants who received study drug in Parts C and D and had EULAR28 evaluated at analysis time points. LOCF was used to impute missing post-baseline values.
Measure: Number; unit: percentage of participants
Groups:
- 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D: Received Placebo, or 1 mg, or 2 mg, or 4 mg LY3009104 in Part A.
  Received 2 mg LY3009104 QD, or BID, or 4 mg LY3009104 QD in Part B.
  Received 4 mg LY3009104 QD in Part C. During Part C, at Weeks 28 and 32, participants who met dose escalation criteria received 8 mg LY3009104 QD for the rest of the Part C.
  Dose escalation criteria: ≥ 6 tender and 6 swollen joints based on the 28-joint count assessments and the clinical judgment of the investigator.
  Received 4 mg LY3009104 QD in Part D.
  MTX was administered orally as background therapy.
Arm/Group | 4 mg LY3009104 QD - Parts C and D | 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D | 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D
Number analyzed (Participants) | 107 | 61 | 31
percentage of participants
  Good Response - Week 76 (n=107, 61, 31) | 64 | 41 | 55
  Moderate Response - Week 76 (n=107, 61, 31) | 27 | 46 | 39
  No Response - Week 76 (n=107, 61, 31) | 8 | 13 | 6
  Good Response - Week 128 (n=79, 47, 18) | 65 | 40 | 56
  Moderate Response - Week 128 (n=79, 47, 18) | 30 | 40 | 28
  No Response - Week 128 (n=79, 47, 18) | 5 | 19 | 17

25. Secondary Outcome: Percentage of Participants Meeting Low Disease Activity and Remission Based on the 28 Diarthrodial Joint Count (DAS28) Baseline Through Weeks 12 and 24
Description: Disease Activity Score (DAS) modified to include 28-joint count (DAS28) consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), CRP [milligrams per liter (mg/L)], and Patient's Global Assessment of Disease Activity using VAS (patient's global VAS). Scores ranged from 1.0-9.4, where lower scores indicated less disease activity. DAS28 scores ≤3.2 are considered as low disease activity, and scores <2.6 are considered as remission. Participants who discontinue before analysis time points are treated as non-responders.
Time Frame: Baseline through Weeks 12 and 24
Population: All randomized participants who received study drug in Parts A and B and had DAS28-CRP evaluated at analysis time points.
Measure: Number; unit: percentage of participants
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 49 | 52 | 52 | 50 | 98
percentage of participants
  Low Disease Activity - Week 12 | 22 | 23 | 48 | 40 | 19
  Remission - Week 12 | 14 | 15 | 37 | 22 | 4
  Low Disease Activity - Week 24 | NA — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore percentage was not calculated. | 31 | 50 | 46 | NA — Participants were not dosed with placebo after Week 12, therefore percentage was not calculated.
  Remission - Week 24 | NA — Participants were not dosed with 1 mg LY3009104 after Week 12, therefore percentage was not calculated. | 15 | 33 | 36 | NA — Participants were not dosed with placebo after Week 12, therefore percentage was not calculated.
Statistical Analysis 1: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.409, Fisher Exact — P-value is for Low Disease Activity - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 2: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.371, Fisher Exact — P-value is for Low Disease Activity - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 3: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact — P-value is for Low Disease Activity - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 4: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.007, Fisher Exact — P-value is for Low Disease Activity - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 5: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.033, Fisher Exact — P-value is for Remission - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 6: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.019, Fisher Exact — P-value is for Remission - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 7: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact — P-value is for Remission - Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 8: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.001, Fisher Exact — P-value is for Remission - Week 12. A priori p-value significance threshold: 2-sided ≤0.10

26. Secondary Outcome: Percentage of Participants Meeting Low Disease Activity and Remission Based on the 28 Diarthrodial Joint Count (DAS28) Baseline Through Weeks 76 and 128
Description: Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consisted of composite score of following variables: tender joint count (TJC28), swollen joint count (SJC28), CRP (mg/L), and Patient's Global Assessment of Disease Activity using VAS (patient's global VAS). Scores ranged from 1.0-9.4, where lower scores indicated less disease activity. DAS28 scores ≤3.2 are considered as low disease activity, and scores <2.6 are considered as remission. Participants who discontinue before analysis time points are treated as non-responders.
Time Frame: Baseline through Weeks 76 and 128
Population: All participants who received study drug in Parts C and D and had DAS28-CRP evaluated at analysis time points.
Measure: Number; unit: percentage of participants
Arm/Group | 4 mg LY3009104 QD - Parts C and D | 4 to 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D | 8 mg LY3009104 QD - Part C and 4 mg LY3009104 QD - Part D
Number analyzed (Participants) | 108 | 61 | 32
percentage of participants
  Low Disease activity - Week 76 (n=108, 61, 32) | 58 | 38 | 44
  Remission - Week 76 (n=108, 61, 32) | 52 | 21 | 22
  Low Disease activity - Week 128 (n=79, 47, 18) | 59 | 36 | 56
  Remission - Week 128 (n=79, 47, 18) | 47 | 26 | 39

27. Secondary Outcome: Mean Change From Baseline Through Week 12 in Duration (Minutes) of Morning Stiffness
Description: The Investigator asked participants about the duration of their morning stiffness (in minutes) in and around the joints and recorded the duration. The Investigator asked the participants about duration of morning stiffness on the day prior to the study visit to capture actual symptoms. If morning stiffness duration was longer than 12 hours (720 minutes), it was truncated to 720 minutes for statistical presentations and analyses.
Time Frame: Baseline, Weeks 4, 8, 12
Population: All randomized participants who received study drug in Part A and had morning stiffness evaluated at analysis time points. LOCF was used to impute missing post-baseline values for Week 12 analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 48 | 51 | 50 | 50 | 97
minutes
  Week 4 (n=47, 50, 50, 50, 94) | -34.1 (70.49) | -27.0 (46.49) | -57.4 (149.00) | -25.5 (126.13) | -22.5 (63.61)
  Week 8 (n=46, 50, 50, 50, 86) | -41.2 (85.45) | -31.1 (45.80) | -67.8 (138.02) | -53.8 (101.76) | -25.5 (67.39)
  Week 12 (n=48, 51, 50, 50, 97) | -49.5 (72.80) | -30.7 (47.41) | -75.0 (142.04) | -62.7 (88.27) | -33.9 (91.79)
Statistical Analysis 1: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.015, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 2: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.073, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 3: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 4: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 12. A priori p-value significance threshold: 2-sided ≤0.10

28. Secondary Outcome: Mean Change From Baseline to Week 12 in Medical Outcomes Study 36-Item Short Form (SF-36) Health Survey Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains (physical functioning, bodily pain, role limitations due to physical problems and also emotional problems, general health, mental health, social functioning and vitality) and 2 component scores (PCS and MCS). The PCS score consisted of physical functioning, bodily pain, role-physical, and general health scales. The MCS score consisted of social functioning, vitality, mental health, and role-emotional scales. Both PCS and MCS range from 0-100 with higher scores indicating better health or functioning.
Time Frame: Baseline, Week 12
Population: All randomized participants who received study drug in Part A and had SF-36 evaluated at analysis time point. LOCF was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 48 | 51 | 51 | 50 | 97
units on a scale
  PCS | 6.66 (8.074) | 4.15 (7.680) | 7.07 (7.378) | 7.00 (9.054) | 3.22 (6.733)
  MCS | 2.54 (11.983) | 1.89 (6.869) | 2.39 (7.898) | 3.03 (10.675) | 0.88 (10.437)
Statistical Analysis 1: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.021, ANCOVA — P-value is for PCS. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 2: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.194, ANCOVA — P-value is for PCS. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 3: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for PCS. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 4: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.012, ANCOVA — P-value is for PCS. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 5: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.449, ANCOVA — P-value is for MCS. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 6: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.578, ANCOVA — P-value is for MCS. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 7: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.140, ANCOVA — P-value is for MCS. A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 8: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.266, ANCOVA — P-value is for MCS. A priori p-value significance threshold: 2-sided ≤0.10

29. Secondary Outcome: Mean Change From Baseline to Week 12 in Brief Pain Inventory Modified Short Form (BPI-sf Modified) Worst-Pain-in-the Past-24-hours Item Score
Description: The BPI-sf modified is a self-administered questionnaire developed for the rapid assessment of pain. The BPI-sf modified provides information on the intensity of pain (the sensory dimension) as well as the degree to which pain interferes with function (the reactive dimension). The questionnaire asks questions about pain relief, pain quality, and the participant's perception of the cause of pain. The BPI-sf modified uses a numeric rating scale from 0 ("No pain") to 10 ("Pain as bad as you can imagine"). Since pain can be quite variable over a day, the BPI-sf modified asked participants to rate their pain at the time of responding to the questionnaire (right now), and also at its worst, least and average over the last 24 hours.
Time Frame: Baseline, Week 12
Population: All randomized participants who received study drug and had BPI-sf worst-pain-in-the past-24-hours item evaluated at Week 12. LOCF was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 48 | 51 | 51 | 50 | 97
units on a scale | -1.35 (2.547) | -0.67 (2.132) | -1.41 (1.813) | -1.54 (2.131) | -0.35 (2.136)
Statistical Analysis 1: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.005, ANCOVA; A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 2: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.135, ANCOVA — A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 3: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 4: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — A priori p-value significance threshold: 2-sided ≤0.10

30. Secondary Outcome: Mean Change From Baseline to Week 12 in Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F) Score
Description: The FACIT-F Scale is a brief 13-item, symptom-specific questionnaire that specifically assesses the participant self-reported severity of fatigue and its impact upon daily activities and functioning. The FACIT-F uses a numeric rating scale of 0 ("Not at all") to 4 ("Very much") for each item to assess fatigue and its impact in the past 7 days. Total scores range from 0 to 52, with higher scores indicating less fatigue.
Time Frame: Baseline, Week 12
Population: All randomized participants who received study drug in Part A and had FACIT-F evaluated at Week 12. LOCF was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 48 | 51 | 51 | 50 | 97
units on a scale | 4.48 (10.492) | 3.80 (9.152) | 4.41 (8.631) | 4.11 (9.971) | 2.02 (8.941)
Statistical Analysis 1: Comparison: 1 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.203, ANCOVA — A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 2: Comparison: 2 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.164, ANCOVA — A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 3: Comparison: 4 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.018, ANCOVA — A priori p-value significance threshold: 2-sided ≤0.10
Statistical Analysis 4: Comparison: 8 mg LY3009104 vs Placebo; Test type: Superiority or Other; p = 0.097, ANCOVA — A priori p-value significance threshold: 2-sided ≤0.10

31. Secondary Outcome: Population Pharmacokinetics (PK): Maximum Concentration at Steady State of Dosing (Cmax,ss) of LY3009104
Time Frame: Baseline through 24 weeks
Population: All randomized participants who received at least 1 dose of LY3009104 with evaluable LY3009104 PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles/Liter (nmol/L)
Groups:
- 2 mg LY3009104: 2 mg LY3009104 administered orally QD for 24 weeks in Parts A and B.
  Participants who received Placebo or 1 mg LY3009104 in Part A were re-randomized at Week 12 to receive 2 mg LY3009104 BID in Part B.
  MTX was administered orally as background therapy.
- 4 mg LY3009104: 4 mg LY3009104 administered orally QD for 24 weeks in Parts A and B.
  Participants who received Placebo or 1 mg LY3009104 in Part A were re-randomized at Week 12 to receive 4 mg LY3009104 QD in Part B.
  MTX was administered orally as background therapy.
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104
Number analyzed (Participants) | 47 | 91 | 91 | 50
nanomoles/Liter (nmol/L) | 36.5 (36.1) | 59.1 (21.3) | 119.0 (20.5) | 241.0 (22.9)

32. Secondary Outcome: Population PK: Area Under the Concentration Curve Versus Time at a Dosing Interval at Steady State (AUCtau,ss) of LY3009104
Time Frame: Baseline through 24 weeks
Population: All randomized participants who received at least 1 dose of LY3009104 with evaluable LY3009104 PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles*hour/Liter (nmol*h/L)
Groups:
- 1mg LY3009104: 1 mg LY3009104 administered orally QD for 12 weeks in Part A. MTX was administered orally as background therapy.
Arm/Group | 1mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104
Number analyzed (Participants) | 47 | 91 | 91 | 50
nanomoles*hour/Liter (nmol*h/L) | 333 (61.7) | 541 (38.0) | 1060 (37.0) | 2190 (45.6)

33. Secondary Outcome: Mean Change From Baseline Through Week 12 in the ENSEMBLE Minimum Data Set 1.0
Time Frame: Baseline, 12 weeks
Population: Zero participants were analyzed. Assessment of ENSEMBLE Minimum Data Set 1.0 was not collected at Week 12 and therefore results are not reported for outcome measure.
Arm/Group | 1 mg LY3009104 | 2 mg LY3009104 | 4 mg LY3009104 | 8 mg LY3009104 | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- 1 mg LY3009104 QD - Part A; 2 mg LY3009104 QD - Part A; 8 mg LY3009104 QD - Part A: Administered orally QD for 12 weeks in Part A.
  MTX was administered orally as background therapy.
- 4 mg LY3009104 QD - Part A: Administered orally QD for 12 weeks in Pat A.
  MTX was administered orally as background therapy.
- 2 mg LY3009104 BID Crossover- Part B: Participants who received Placebo or 1 mg LY3009104 in Part A were re-randomized at Week 12 to receive 2 mg LY3009104 BID in Part B.
  MTX was administered orally as background therapy.
- 4 mg LY3009104 QD Crossover- Part B: Participants who received Placebo or 1 mg LY3009104 in Part A were re-randomized at Week 12 to receive 4 mg LY3009104 QD in Part B.
  MTX was administered orally as background therapy.
- 2 mg LY3009104 QD - Part B: Participants who received 2 mg LY3009104 QD in Part A continued to receive 2 mg LY3009104 QD in Part B.
  MTX was administered orally as background therapy.
- 4 mg LY3009104 QD - Part B: Participants who received 4 mg LY3009104 QD in Part A continued to receive 4 mg LY3009104 QD in Part B.
  MTX was administered orally as background therapy.
- 8 mg LY3009104 QD - Part B: Participants who received 8 mg LY3009104 QD in Part A continued to receive 8 mg LY3009104 QD in Part B.
  MTX was administered orally as background therapy.
- 4 mg LY3009104 QD - Part C: Participants who received 2 mg LY3009104 QD or BID in Part B were re-assigned at Week 24 to 4 mg LY3009104 QD in Part C.
  Participants who received 4 mg LY3009104 QD in Part B continued to receive 4 mg LY3009104 QD in Part C.
  MTX was administered orally as background therapy.
- 4 to 8 mg LY3009104 QD Pre-Rescue - Part C: Participants who received 2 mg LY3009104 QD or BID in Part B were re-assigned at Week 24 to 4 mg LY3009104 QD in Part C.
  Participants who received 4 mg LY3009104 QD in Part B continued to receive 4 mg LY3009104 QD in Part C.
  During Part C, at Weeks 28 and 32, participants who met dose escalation criteria received 8 mg LY3009104 QD (rescue treatment) for the rest of the Part C.
  MTX was administered orally as background therapy.
  Adverse events were collected from Week 24 until predose of 8 mg LY3009104 QD.
- 4 to 8 mg LY3009104 QD Post-Rescue - Part C: Participants who received 2 mg LY3009104 QD or BID in Part B were re-assigned at Week 24 to 4 mg LY3009104 QD in Part C.
  Participants who received 4 mg LY3009104 QD in Part B continued to receive 4 mg LY3009104 QD in Part C.
  During Part C, at Weeks 28 and 32, participants who met dose escalation criteria received 8 mg LY3009104 QD (rescue treatment) for the rest of the Part C.
  MTX was administered orally as background therapy.
  Adverse events were collected from predose of 8 mg LY3009104 QD until Week 76.
- 8 mg LY3009104 QD - Part C: Participants who received 8 mg LY3009104 QD in Part B remained on 8 mg LY3009104 QD in Part C.
  MTX was administered orally as background therapy.
- 4 mg LY3009104 QD - Part D: Participants who received 4 mg LY3009104 QD in Part C continued to receive 4 mg LY3009104 QD in Part D.
  MTX was administered orally as background therapy.
- 4 mg LY3009104 QD (4 to 8 mg Rescue)- Part D: Participants who received 8 mg LY3009104 QD rescue treatment in Part C received 4 mg LY3009104 QD in Part D.
  MTX was administered orally as background therapy.
- 8/4 mg LY3009104 QD - Part D: Participants who received 8 mg LY3009104 QD in Part C received 4 mg LY3009104 QD in Part D.
  MTX was administered orally as background therapy.
- Follow-Up: Up to 28 days post the last dose of study drug.
  MTX was administered orally as background therapy.
Arm/Group | 1 mg LY3009104 QD - Part A | 2 mg LY3009104 QD - Part A | 4 mg LY3009104 QD - Part A | 8 mg LY3009104 QD - Part A | Placebo QD - Part A | 2 mg LY3009104 BID Crossover- Part B | 4 mg LY3009104 QD Crossover- Part B | 2 mg LY3009104 QD - Part B | 4 mg LY3009104 QD - Part B | 8 mg LY3009104 QD - Part B | 4 mg LY3009104 QD - Part C | 4 to 8 mg LY3009104 QD Pre-Rescue - Part C | 4 to 8 mg LY3009104 QD Post-Rescue - Part C | 8 mg LY3009104 QD - Part C | 4 mg LY3009104 QD - Part D | 4 mg LY3009104 QD (4 to 8 mg Rescue)- Part D | 8/4 mg LY3009104 QD - Part D | Follow-Up
Serious Adverse Events (participants affected / at risk) | 0/49 | 3/52 | 2/52 | 1/50 | 3/98 | 2/63 | 1/63 | 0/51 | 0/50 | 3/49 | 16/108 | 1/61 | 6/61 | 6/32 | 5/79 | 3/47 | 0/18 | 2/159
Other Adverse Events (participants affected / at risk) | 15/49 | 13/52 | 13/52 | 15/50 | 18/98 | 15/63 | 10/63 | 12/51 | 10/50 | 18/49 | 35/108 | 7/61 | 25/61 | 16/32 | 24/79 | 13/47 | 10/18 | 5/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1 mg LY3009104 QD - Part A (N=49) | 2 mg LY3009104 QD - Part A (N=52) | 4 mg LY3009104 QD - Part A (N=52) | 8 mg LY3009104 QD - Part A (N=50) | Placebo QD - Part A (N=98) | 2 mg LY3009104 BID Crossover- Part B (N=63) | 4 mg LY3009104 QD Crossover- Part B (N=63) | 2 mg LY3009104 QD - Part B (N=51) | 4 mg LY3009104 QD - Part B (N=50) | 8 mg LY3009104 QD - Part B (N=49) | 4 mg LY3009104 QD - Part C (N=108) | 4 to 8 mg LY3009104 QD Pre-Rescue - Part C (N=61) | 4 to 8 mg LY3009104 QD Post-Rescue - Part C (N=61) | 8 mg LY3009104 QD - Part C (N=32) | 4 mg LY3009104 QD - Part D (N=79) | 4 mg LY3009104 QD (4 to 8 mg Rescue)- Part D (N=47) | 8/4 mg LY3009104 QD - Part D (N=18) | Follow-Up (N=159)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute hepatitis b (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/42 (0) | 0/44 (0) | 0/37 (0) | 0/41 (0) | 0/85 (0) | 0/56 (0) | 0/54 (0) | 0/43 (0) | 0/35 (0) | 0/40 (0) | 0/87 (0) | 0/52 (0) | 0/52 (0) | 0/28 (0) | 0/62 (0) | 0/40 (0) | 0/17 (0) | 1/130 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/42 (0) | 0/44 (0) | 0/37 (0) | 0/41 (0) | 0/85 (0) | 0/56 (0) | 0/54 (0) | 0/43 (0) | 0/35 (0) | 0/40 (0) | 0/87 (0) | 0/52 (0) | 1/52 (1) | 0/28 (0) | 0/62 (0) | 0/40 (0) | 0/17 (0) | 0/130 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg LY3009104 QD - Part A (N=49) | 2 mg LY3009104 QD - Part A (N=52) | 4 mg LY3009104 QD - Part A (N=52) | 8 mg LY3009104 QD - Part A (N=50) | Placebo QD - Part A (N=98) | 2 mg LY3009104 BID Crossover- Part B (N=63) | 4 mg LY3009104 QD Crossover- Part B (N=63) | 2 mg LY3009104 QD - Part B (N=51) | 4 mg LY3009104 QD - Part B (N=50) | 8 mg LY3009104 QD - Part B (N=49) | 4 mg LY3009104 QD - Part C (N=108) | 4 to 8 mg LY3009104 QD Pre-Rescue - Part C (N=61) | 4 to 8 mg LY3009104 QD Post-Rescue - Part C (N=61) | 8 mg LY3009104 QD - Part C (N=32) | 4 mg LY3009104 QD - Part D (N=79) | 4 mg LY3009104 QD (4 to 8 mg Rescue)- Part D (N=47) | 8/4 mg LY3009104 QD - Part D (N=18) | Follow-Up (N=159)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acquired oesophageal web (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 9 (9) | 0 (0) | 3 (3) | 5 (5) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 7 (9) | 2 (2) | 2 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 9 (10) | 1 (1) | 6 (8) | 1 (1) | 3 (5) | 2 (3) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 12 (15) | 1 (1) | 5 (6) | 3 (3) | 3 (4) | 1 (1) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Spinal laminectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days